CLINICAL TRIAL: NCT06740903
Title: Comparison of Dexmedetomidine & Lignocaine Infusion on Perioperative Hemodynamics, Postoperative Analgesia & Recovery of Postoperative Gastrointestinal Function in Patients for Laparoscopic Cholecystectomy
Brief Title: Evaluating Perioperative Outcomes: Dexmedetomidine vs Lignocaine in Laparoscopic Chlolecystectomy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sahiwal medical college sahiwal (Other Government)
Collaborators: Department of medical education (Unknown)
Responsible Party: Principal Investigator, Talal Shahid, Resident Anaesthetist, Sahiwal medical college sahiwal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 84/IRB/SLMC/SWL
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hemodynamics Instability; Post Operative Pain; Gastrointestinal Dysfunction; Cholecystitis
MeSH Terms: conditions — Pain, Postoperative; Cholecystitis | interventions — Dexmedetomidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine infusion (Experimental): inj dexmedetomidine infusion @ 0.2-0.4 μg/kg/h
  Interventions: Drug: inj. dexmedetomidine infusion @ 0.2-0.4 μg/kg/h
- Lignocaine infusion (Experimental): inj.lignocaine infusion @1-2 mg/kg/h
  Interventions: Drug: inj. lignocaine infusion @1-2 mg/kg/h

INTERVENTIONS:
Drug: inj. dexmedetomidine infusion @ 0.2-0.4 μg/kg/h — Anesthesia induction will be done by doing pre-oxygenation for 3 minutes with 100% oxygen, propofol 2-2.5 mg/kg intravenous (IV) and nalbuphine 0.1mg/kg intravenous (IV). Tracheal intubation will be facilitated by succinylcholine 1.5 mg/kg IV. Anaesthesia will be maintained with isoflurane 0.6 mac, 60% nitrous oxide, 40% oxygen, atracurium 0.5mg/kg bolus followed by 0.15mg/kg maintenance dose every 30 mints until completion of surgery. Patients Intraoperative monitoring will include electrocardiogram leads II and V5, non-invasive blood pressure at 5 min intervals, oxygen saturation, end-tidal carbon dioxide and nasopharyngeal temperature. Patients will be ventilated by intermittent positive pressure ventilation using a circle system to maintain normocapnia. In group A, patients will be given inj. dexmedetomidine infusion @ 0.2-0.4 μg/kg/h intraoperatively
  Other Names: Precedex
  Arms: Dexmedetomidine infusion
Drug: inj. lignocaine infusion @1-2 mg/kg/h — Anesthesia induction will be done by doing pre-oxygenation for 3 minutes with 100% oxygen, propofol 2-2.5 mg/kg intravenous (IV) and nalbuphine 0.1mg/kg intravenous (IV). Tracheal intubation will be facilitated by succinylcholine 1.5 mg/kg IV. Anaesthesia will be maintained with isoflurane 0.6 mac, 60% nitrous oxide, 40% oxygen, atracurium 0.5mg/kg bolus followed by 0.15mg/kg maintenance dose every 30 mints until completion of surgery. Patients Intraoperative monitoring will include electrocardiogram leads II and V5, non-invasive blood pressure at 5 min intervals, oxygen saturation, end-tidal carbon dioxide and nasopharyngeal temperature. Patients will be ventilated by intermittent positive pressure ventilation using a circle system to maintain normocapnia. In group A, patients will be given inj. lignocaine infusion @ 1-2 mg/kg/h intraoperatively
  Other Names: Xylocaine
  Arms: Lignocaine infusion

SUMMARY:
Nowadays laparoscopic surgery is the first choice for many surgeries. Such surgeries have revolutionized the surgical practice and has markedly reduced the incidence of intraoperative and postoperative complications. To minimize these side effects associated with the use of opioids, various methods have been adopted. Recently, different trials have highlighted the possible role of dexmedetomidine and lignocaine in providing postoperative analgesia and attenuating hemodynamic response. Literature showed conflicting results regarding both these drugs. So, we want to find the evidence for local setting. This Randomized Controlled Trial will be done at Department of Anesthesia, Sahiwal teaching hospital, Sahiwal for 12 months. Sample size of 140 cases; 70 cases in each group will be included through non-probability consecutive sampling. Then patients will be divided in two groups by using computer generated random number table. In group A, patients will be given dexmedetomidine infusion. In group B, patients will be given lignocaine infusion. All anesthesia procedures will be done by researcher. Heart rate and mean arterial pressure will be assessed before induction of anesthesia, after every 10 mins every 30 mins till completion of surgery. Total operative time will be noted. After procedure, patients will be assessed for postoperative pain score. when pain will be ≥4 on visual analogue scale rescue analgesia will be given and time will be noted. Total duration from time of surgery till need for rescue analgesia will be noted. Duration of postoperative analgesia opioid consumption /24 hrs.) will be presented by using mean± SD.

DETAILED DESCRIPTION:
After approval from hospital ethical committee and obtaining informed written consent from every patient, patient fulfilling the criteria of inclusion. All patients will be categorized into two different groups using computer generated random number table. Demographic information (name, age, gender, weight, ASA) will be noted. All patients will undergo a preoperative assessment on the day before surgery. They will be pre-medicated with oral midazolam 0.05 mg/kg 2 h before surgery. Anesthesia induction will be done by doing pre-oxygenation for 3 minutes with 100% oxygen, propofol 2-2.5 mg/kg intravenous (IV) and nalbuphine 0.1mg/kg intravenous (IV). Tracheal intubation will be facilitated by succinylcholine 1.5 mg/kg IV. Anaesthesia will be maintained with isoflurane 0.6 mac, 60% nitrous oxide, 40% oxygen, atracurium 0.5mg/kg bolus followed by 0.15mg/kg maintenance dose every 30 mints until completion of surgery. Patients Intraoperative monitoring will include electrocardiogram leads II and V5, non-invasive blood pressure at 5 min intervals, oxygen saturation, end-tidal carbon dioxide and nasopharyngeal temperature. Patients will be ventilated by intermittent positive pressure ventilation using a circle system to maintain normocapnia. In group A, patients will be given inj. dexmedetomidine infusion @ 0.2-0.4 μg/kg/h intraoperatively. In group B, patients will be given inj. lignocaine infusion @1-2 mg/kg/h intraoperatively. All anesthesia procedures will be done by researcher under supervision of senior consultant anesthesiologist having at least 4years residency experience. The person who will prepare the study drugs will not participate in the data collection procedure. Heart rate and mean arterial pressure will be assessed before induction of anesthesia, then at 5, 10, 20,30, and every 30 minutes till the completion of surgery. Hypotension (MAP <20% of the baseline or <65 mmHg) will be treated with infusion of normal saline and if required injection phenylephrine boluses IV. Bradycardia (HR <40 beats/min) will be treated with IV atropine 40 µg/kg bolus in both intraoperative and post-operative period. All patients will receive paracetamol 15 mg/kg IV and ondansetron 0.1 mg/kg IV ½ hour before the completion of surgery. At the end of surgery, residual neuromuscular block will be antagonized with 0.05mg/kg of neostigmine and glycopyrrolate IV. Tracheal extubation will be performed on meeting the standard criteria for extubating. Total operative time will be noted. After procedure, patients will be shifted in intensive care unit and will be followed-up there for 24 hours. Patients will be assessed for postoperative pain score. when pain will be ≥4 on visual analogue scale rescue analgesia will be given and time will be noted. Total duration from time of surgery till need for rescue analgesia will be noted (as per operational definition). Total opioid consumption /24 hrs. will be noted along with nausea and vomiting. Recovery of postop gastrointestinal function will be assessed using 5 point I-FEED scale at 6, 12, and 24 hours postoperatively. All the information will be recorded on proforma (attached).

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age 20-70 years
2. Both gender
3. Laparoscopic cholecystectomy under general Anaesthesia
4. ASA I-II.

Exclusion Criteria:

* Emergency surgery
* Patients with history of allergic reaction to trial drugs
* Patients with cardiovascular disease, sickle cell disease, psychiatric disorder, peripheral vascular disease, and neurological diseases (on medical record)
* Anemia
* Patient on TCA or Beta blocker drugs.
* Uncontrolled hypertension (P≥160/100 mmHg)
* Uncontrolled diabetes mellitus
* Obesity BMI > 35

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-08-06 (Estimated); Study Completion 2025-09-06 (Estimated)

PRIMARY OUTCOMES:
HR | heart beats per minute (bpm) before induction of anesthesia, then 5, 10, 20,30, 60,90,120 minutes of anesthesia
  heart rate of the patient
MAP | it will be measured in terms of mmHg before induction of anesthesia, after 5, 10, 20,30, 60,90,120 minutes of anesthesia on ECG monitor
  Mean Arterial Pressure
Post-op Pain | it will be assessed in terms of minuTotal duration from time of surgery till need for rescue analgesia will be noted.
  Post Operative Analgesia

SECONDARY OUTCOMES:
Post-op GIT Functions | Recovery of postop gastrointestinal function will be assessed using 5 point I-FEED scale at 6, 12, and 24 hours postoperatively
  Post-operative GIT Functions by I-FEED Scale

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Riaz, MD, Study Director — Sahiwal Teaching Hospital, Sahiwal
Locations (1):
- Sahiwal Medical College Sahiwal, Sahiwal, Punjab Province, Pakistan